CLINICAL TRIAL: NCT03254602
Title: Intense Therapeutic Ultrasound for the Treatment of Chronic Plantar Fasciitis Musculoskeletal Pain Reduction
Brief Title: Intense Therapeutic Ultrasound for the Treatment of Chronic Plantar Fasciitis
Acronym: ITU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Foot and Ankle Foundation (Other)
Collaborators: Guided Therapy Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160753
Record Dates: First submitted 2017-08-14; First posted 2017-08-18 (Actual); Results first posted 2017-11-17 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-10

CONDITIONS: Plantar Fasciitis, Chronic
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intense Therapeutic Ultrasound Treatment (Experimental): Intense Therapeutic Ultrasound treatment applied along the length and width of the proximal Plantar Fascia. 1000 - 5 Joule pulses were applied twice, four weeks apart.
  Interventions: Device: Intense Therapeutic Ultrasound Treatment

INTERVENTIONS:
Device: Intense Therapeutic Ultrasound Treatment
  Other Names: Guided Therapy Systems, Ardent Sound, GTS, ITU; Actisound

SUMMARY:
A clinical trial evaluating the effectiveness, safety and patient tolerance for the use of Intense Therapeutic Ultrasound (ITU) for chronic, Plantar Fasciitis musculoskeletal tissue pain reduction began in August 2016 and was completed in April 2017. The clinical setting: University Foot and Ankle Institute, Santa Monica, California, USA; Single-Blinded, pivotal study for chronic plantar fasciitis.

DETAILED DESCRIPTION:
Intense Therapeutic Ultrasound (ITU) is an established ultrasound based therapy in which sound waves are concentrated and focused into selected musculoskeletal tissue, to produce selective thermal coagulative changes over a small controlled area while leaving the surrounding tissue unaffected. These coagulative changes are known to begin the body's tissue response cascade and promote collagen generation in the targeted anatomy resulting in pain reduction.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Pain (>90 days) from previously diagnosed Plantar Fasciitis, where "Standard of Care" regimens failed to relief pain in the affected anatomy.
* No History of surgery to the affected anatomy.
* No alternative treatment procedures within the last 90 days.
* Age: 18 - 85, depending on the study.
* Unilateral Pain
* Willingness to complete treatment and post treatment regimen as described.
* Patients who have provided written and verbal informed consent.

Exclusion Criteria:

* Patients currently enrolled in any other non-conservative, device, or Investigational New Drug clinical trial, or who have participated in a clinical study involving the Plantar Fascia, thirty days prior to study initiation;
* Patients who have participated in any other clinical study involving an investigational product 30 days prior to enrollment that, in the opinion of the Principal Investigator, could affect the outcome of this study;
* Patients who have received previous treatment in the symptomatic limb (not including conservative treatment);
* At the Principal Investigator's discretion, any patient that should be excluded based on their current condition or medical history.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bob Baravarian, DPM, Principal Investigator — University Foot and Ankle Foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White WM, Makin IR, Barthe PG, Slayton MH, Gliklich RE. Selective creation of thermal injury zones in the superficial musculoaponeurotic system using intense ultrasound therapy: a new target for noninvasive facial rejuvenation. Arch Facial Plast Surg. 2007 Jan-Feb;9(1):22-9. doi: 10.1001/archfaci.9.1.22. PMID 17224484
- [Background] Alam M, White LE, Martin N, Witherspoon J, Yoo S, West DP. Ultrasound tightening of facial and neck skin: a rater-blinded prospective cohort study. J Am Acad Dermatol. 2010 Feb;62(2):262-9. doi: 10.1016/j.jaad.2009.06.039. PMID 20115948
- [Background] Gliklich RE, White WM, Slayton MH, Barthe PG, Makin IR. Clinical pilot study of intense ultrasound therapy to deep dermal facial skin and subcutaneous tissues. Arch Facial Plast Surg. 2007 Mar-Apr;9(2):88-95. doi: 10.1001/archfaci.9.2.88. PMID 17372061
- [Background] Laubach HJ, Makin IR, Barthe PG, Slayton MH, Manstein D. Intense focused ultrasound: evaluation of a new treatment modality for precise microcoagulation within the skin. Dermatol Surg. 2008 May;34(5):727-34. doi: 10.1111/j.1524-4725.2008.34196.x. PMID 18429926
- [Background] Molloy T, Wang Y, Murrell G. The roles of growth factors in tendon and ligament healing. Sports Med. 2003;33(5):381-94. doi: 10.2165/00007256-200333050-00004. PMID 12696985
- [Background] Landorf KB, Keenan AM, Herbert RD. Effectiveness of foot orthoses to treat plantar fasciitis: a randomized trial. Arch Intern Med. 2006 Jun 26;166(12):1305-10. doi: 10.1001/archinte.166.12.1305. PMID 16801514

RESULTS

PARTICIPANT FLOW:
Groups:
- Intense Therapeutic Ultrasound Treatment: Intense Therapeutic Ultrasound treatment applied along the length and width of the proximal Plantar Fascia. 1000 - 5 Joule pulses were applied twice, four weeks apart.
  Intense Therapeutic Ultrasound Treatment
Period: Overall Study
Arm/Group | Intense Therapeutic Ultrasound Treatment
Started | 33
Completed | 29
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Intense Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants] — Patient Age at time of first treatment
  Participants
    <=18 years | 0
    Between 18 and 65 years | 30
    >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 56 [31 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33
Patients with Chronic Plantar Fasciitis where Standard of Care Therapy failed to Reduce Pain [Count of Participants; unit: Participants] | 33

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Pain Via the Universal Visual Analog Scale: Pass Criteria = at Least 25% Pain Reduction
Description: Patient Reported Pain Reduction meeting or exceeding 25% using the Universal Visual Analog Scale. The Universal Visual Analog Scale is a 10 Point pain scale, where 0 = No Pain, 1 = slight Pain and 10 = the patient's worst imaginable pain. Ratings of 2 to 9 describe pain increases of 10%/Rating. For this measure a reduction of 25% on the Universal Visual Analog Scale is considered meeting the Pain Reduction Criteria. Lower Scale numbers compared to reported baseline ratings equates to pain reduction.
Time Frame: At 12 weeks after the first treatment
Population: Patients receiving 2 Intense Therapeutic Ultrasound Treatments, beginning 12 Weeks ago.
Measure: Number; unit: Percent of Patients meeting criteria
Arm/Group | Intense Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 29
Percent of Patients meeting criteria | 86

2. Secondary Outcome: Ultrasound Changes
Description: Diagnostic Ultrasound Changes: Hypoechoic Lesion Volume Reduction following 2 Intense Therapeutic Ultrasound Treatments
Time Frame: At 12 Weeks after the first treatment
Population: Patients receiving 2 Intense Therapeutic Ultrasound Treatments - Average % Volume Reduction of Hypoechoic Plantar Fascia Lesions
Measure: Mean (Full Range); unit: percentage of Lesion Size Reduction
Arm/Group | Intense Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 26
percentage of Lesion Size Reduction | 56 [0 to 100]

3. Secondary Outcome: Percentage of Change of Pain and Hypoechoic Lesion Volume Compared to Baseline
Description: Compare percentage of Mean changes in pain via the Patient Reported Universal Visual Analog Scale compared to Mean Patient Reported Baseline Pain Scores and percentage of Mean change of Plantar Fascia Hypoechoic Lesion Volume compared to mean baseline Hypoechoic lesion volume following two Intense Therapeutic Ultrasound Treatments, using Diagnostic Ultrasound Images. For Plantar Fascia Hypoechoic Lesion Volume, each lesion volume was calculated using: (4/3) π x R1 x R2 x R3, where r = Radius of each measurement: Lesion Length(1), width(2) and depth(3)
Time Frame: At 12 Weeks after the first treatment
Population: Patients receiving 2 Intense Therapeutic Ultrasound treatments beginning 12 weeks ago
Measure: Mean (Full Range); unit: percentage of Change
Arm/Group | Intense Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 26
percentage of Change
  Mean % PF Pain Change | -54 [-100 to 100]
  Mean % Change in PF Hypoechoic Lesion Volume | -56 [-100 to 100]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Any patient reported event occurring after the first treatment.
Arm/Group | Intense Therapeutic Ultrasound Treatment
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
Bias was mitigated as much as possible within the protocol by way of the blinding throughout the layers of patients and personnel involved in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT03254602/ICF_000.pdf
  • Study Protocol (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03254602/Prot_001.pdf
  • Statistical Analysis Plan (2016-05-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT03254602/SAP_002.pdf